CLINICAL TRIAL: NCT03560635
Title: Feasibility and Preliminary Efficacy of a Reverse Diet as a Novel Weight Loss Maintenance Strategy for Weight-Reduced Adults With Overweight/Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-1726
Record Dates: First submitted 2018-05-21; First posted 2018-06-18 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity; Weight Loss Maintenance; Dietary Habits
Keywords: weight loss maintenance; reverse diet; body composition; metabolic rate; dietary adherence; resting energy expenditure; weight loss; weight regain
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants randomized to the CON condition will be informed of their estimated weight maintenance calorie needs (determined by multiplying their resting energy expenditure (REE) obtained from indirect calorimetry by an appropriate activity factor and advised to adhere to this calorie target, as is standard weight maintenance advice. Participants will be provided with a food scale and calorie tracking options and instructed on the importance of high adherence to the diet protocol.
  Interventions: Behavioral: Weight Loss Maintenance (Control vs. Reverse Diet)
- Reverse Diet (Experimental): Participants randomized to the reverse diet condition will receive specific caloric intake goals. The initial caloric goal will be set at 2-3% above the level participants ended their weight loss diet at (via self-report). Participants' caloric goals will increase at a rate of 2-3% per week. Participants will be provided with a food scale and calorie tracking options and instructed on the importance of high adherence to the reverse diet protocol.
  Interventions: Behavioral: Weight Loss Maintenance (Control vs. Reverse Diet)

INTERVENTIONS:
Behavioral: Weight Loss Maintenance (Control vs. Reverse Diet) — Participants in both groups will receive a 12-week comprehensive, individually delivered behavioral weight loss maintenance intervention, adapted from the Diabetes Prevention Program (DPP) Post-CORE program. This program focuses on utilization of tools and strategies to maintain a healthy lifestyle and prevent weight regain, and is therefore most appropriate for the weight-reduced population we will enroll. While the DPP Post-CORE program includes 15 sessions delivered over 15-months, we will deliver sessions #1-12 and 15 over a 12-week period. Content for sessions 13 and 14 from the DPP Post-CORE curriculum focus specifically on Type 2 Diabetes Mellitus and Heart Disease. The informational handouts will be provided to participants, but not specifically covered in weekly meetings. Groups will differ only in specific caloric prescriptions (described in the Arms section).

SUMMARY:
The purpose of this project is to test, for the first time, a reverse diet in adults with current or prior overweight/obesity (Ow/Ob). Weight-reduced adults with current or prior Ow/Ob will be randomized to a reverse diet or "standard care" control (CON) intervention for 12 weeks. Eligible participants will have lost >10% body mass. The reverse diet group will receive personalized caloric intake goals, increasing 2-3%/week. The CON group will receive standard weight maintenance recommendations with matched contact. At baseline and week 12, resting energy expenditure (REE), body mass and composition, subjective appetite, and food intake behaviors will be evaluated. In addition to the pre- and post-intervention measures, body mass and adherence to reverse diet will be monitored weekly.

ELIGIBILITY:
Inclusion Criteria:

* All ethnic groups and both genders
* Age: 21-70 years
* BMI: 18.5-40 kg/m2
* Weight loss of >10% body mass achieved within 4 weeks of enrollment in study.

Exclusion Criteria:

* Uncontrolled cardio metabolic disease such as: cardiovascular disease (CVD), diabetes mellitus, hypertension (defined as: systolic blood pressure >160 mmHg or diastolic blood pressure >100mmHg, as measured during the screening visit with participants seated quietly, following established guidelines), renal disease (e.g. chronic kidney disease, polycystic kidney disease, nephritis, etc.), hepatic disease (e.g. cirrhosis, liver failure, fatty liver, jaundice, etc.), untreated thyroid disease (e.g. Grave's disease, Hashimoto's disorder, goiters, thyroid cancers, etc.), or any other medical condition affecting weight or energy metabolism. Participants who are deemed ineligible based upon uncontrolled hypertension criteria will be referred to their primary care physicians for treatment. If these conditions become controlled they will be allowed to be re-evaluated for inclusion in the current trial.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Significant gastrointestinal disorders including: inflammatory bowel disease requiring treatment within the past year, chronic malabsorptive conditions, chronic diarrhea, or active gallbladder disease.
* Use of pharmacotherapy agents to achieve weight loss prior to study enrollment.
* Current treatment with medications known to significantly affect appetite, weight, energy metabolism, energy intake or energy expenditure. (e.g. systemic corticosteroids, appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants).
* History of surgical or endoscopic procedure for weight loss at any time (e.g. gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve, intragastric balloons, aspiration therapy, etc); history of extensive bowel resection for other reasons.
* Currently pregnant, lactating or less than 6 months post-partum.
* Planning to become pregnant during study enrollment period
* Self-report of alcohol or substance abuse within the past 12 months.
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder, or score >20 on the EATS-26. Participants with a score >20 on the EATS-26 will be referred to their primary care physician for further evaluation.
* Major psychiatric disorder (e.g. diagnosis of schizophrenia, bipolar disorder, or other psychotic disorders).
* Current severe depression or history of severe depression within the previous year (based on reported history, study physician examination findings, and/or a score >21 on the CES-D). Participants meeting any of these criteria will be referred to their primary care physician and/or the emergency department (based upon study physician determined level of severity).
* Currently participating in or planning to participate in any formal weight loss programs or clinical trials.
* Other medical, psychiatric, or behavioral limitations that may interfere with participation (as determined by study physician).
* Unable or unwilling to undergo study procedures

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Adherence to the prescribed diet | 12 weeks
  Self-reported caloric intake compared to prescribed caloric intake
Adherence to the prescribed diet | 12 weeks
  Evaluated via mathematical model based on change in body mass and composition.
Enrollment Success | 9 months
  The investigators will assess whether they are able to enroll 24 participants meeting study inclusion/exclusion criteria over a 9-month recruitment window. If enrollment is <24, the investigators will determine barriers to enrollment and re-evaluate the study design and/or recruitment strategies. The investigators will also assess participation rate (number approached versus enrolled), reasons potential participants decline enrollment, and ability to meet demographic goals for the larger trial (approximately equal men and women, ≥33% racial and ethnic minorities).
Attrition Rate | 12 Months
  The investigators will assess the participant drop-out rate and reasons for attrition over the 12-week study, determine reasons for drop-outs and examine whether drop-out rates differ between intervention arms.

SECONDARY OUTCOMES:
Changes in Body Mass | Measured weekly throughout the 12-week trial.
  Measured via calibrated digital scale.
Changes in Body Composition | At baseline and post intervention (Week 12).
  Measured via Dual-energy X-ray absorptiometry (DXA) scan
Changes in Resting Energy Expenditure | At baseline and post intervention (Week 12).
  Measured via standard indirect calorimetry with ventilated hood technique
Dietary Adherence | Measured weekly throughout the 12-week trial.
  Evaluated via self-report using a measure created by researchers:
  * "How adherent were you to the prescribed diet over the past week?",
  * measured by self-report from 1 (not at all) to 10 (very much so),
  * higher scores indicate higher dietary adherence
Effort | Weekly, throughout the 12-Week Trial
  Measure created by researchers:
  * "How hard was it to adhere to the prescribed diet over the last week?"
  * measured by self-report from 1(very easy) to 10 (very difficult)
  * higher scores indicate more expended effort
Self-Efficacy | Weekly, throughout the 12-Week Trial
  Measure created by researchers:
  * "How likely do you feel you can adhere to the prescribed diet for the next week?"
  * measured by self-report from 1(not at all likely) to 10 (very likely)
  * higher scores indicate higher self-efficacy
Changes in Food-Related Behaviors | At baseline and post intervention (Week 12).
  Evaluated via Three-Factor Eating Questionnaire, which is divided into three subscales:
  * Factor One: Dietary Restraint (higher scores indicate higher levels of restrained eating)
  * Factor Two: Dis-inhibition of Control (higher scores indicate higher levels of disinhibited eating)
  * Factor Three: Susceptibility to Hunger (higher scores indicate higher levels of predisposition to hunger)
Changes in Food-Related Behaviors | At baseline and post intervention (Week 12).
  Evaluated via the Weight Efficacy Lifestyle Questionnaire, which is divided into five subscales:
  * Negative Emotions
  * Availability
  * Social Pressure
  * Physical Discomfort
  * Positive Activities

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Halliday, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Denver, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No